CLINICAL TRIAL: NCT07397949
Title: A Randomized Noninferiority Trial Comparing Rebamipide and Diquafosol for Perioperative Dry Eye Management in Cataract Surgery
Brief Title: Rebamipide Versus Diquafosol for Perioperative Dry Eye in Cataract Surgery
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Dong Hui Lim, Associate Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RVK-25-I01
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Dry Eye Disease (DED); Cataract
MeSH Terms: conditions — Dry Eye Syndromes; Cataract | interventions — rebamipide; Ophthalmic Solutions; diquafosol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rebamipide Group (Experimental): Participants receive topical rebamipide 2% ophthalmic solution administered four times daily to the surgical eye, starting 1 month before cataract surgery and continuing for 3 months postoperatively.
  Interventions: Drug: Rebamipide 2% ophthalmic solution
- Diquafosol Group (Active Comparator): Participants receive topical diquafosol 3% ophthalmic solution administered four times daily to the surgical eye, starting 1 month before cataract surgery and continuing for 3 months postoperatively.
  Interventions: Drug: Diquafosol 3% ophthalmic solution

INTERVENTIONS:
Drug: Rebamipide 2% ophthalmic solution — Topical administration to the surgical eye, four times daily.
  Arms: Rebamipide Group
Drug: Diquafosol 3% ophthalmic solution — Topical administration to the surgical eye, four times daily.
  Arms: Diquafosol Group

SUMMARY:
This clinical trial is designed to compare two commonly used eye drop treatments for dry eye disease in patients undergoing cataract surgery.

Dry eye disease is common in people who need cataract surgery and may worsen before or after surgery, causing eye discomfort, blurred vision, and unstable vision. Proper management of dry eye before and after surgery may help improve eye comfort and the accuracy of vision outcomes.

In this study, patients with mild to moderate dry eye disease who are scheduled for cataract surgery will be randomly assigned to receive one of two treatments:

Rebamipide eye drops, or

Diquafosol eye drops

Participants will begin using the assigned eye drops one month before cataract surgery and continue treatment for three months after surgery. The eye drops will be used only in the eye undergoing surgery.

Researchers will examine whether one treatment is as effective as the other in improving tear film stability and reducing dry eye symptoms around the time of cataract surgery. Eye examinations and questionnaires will be performed before surgery, on the day of surgery, and during follow-up visits after surgery.

The information gained from this study may help doctors choose the most appropriate treatment for managing dry eye disease in patients undergoing cataract surgery.

DETAILED DESCRIPTION:
Dry eye disease (DED) is frequently observed in patients undergoing cataract surgery and may be exacerbated by surgical trauma, postoperative inflammation, and disruption of corneal innervation. Worsening of dry eye symptoms during the perioperative period can negatively affect patient comfort, tear film stability, and visual outcomes after surgery. Therefore, effective perioperative management of dry eye disease is an important component of cataract surgery care.

This study is a prospective, randomized, parallel-group, investigator-initiated clinical trial designed to compare the efficacy of rebamipide 2% ophthalmic solution and diquafosol 3% ophthalmic solution for perioperative management of dry eye disease in patients undergoing cataract surgery.

Eligible adult patients with mild to moderate dry eye disease who are scheduled for unilateral cataract surgery will be randomly assigned in a 1:1 ratio to one of two treatment groups. Participants will receive either rebamipide or diquafosol eye drops administered to the surgical eye, starting one month before cataract surgery and continuing for three months postoperatively. Standard postoperative medications for cataract surgery will be administered according to routine clinical practice.

The primary outcome measure is the change in tear film breakup time (TBUT) from baseline to the postoperative period. Secondary outcome measures include changes in corneal staining grade, patient-reported symptoms assessed using the Ocular Surface Disease Index (OSDI), tear secretion measured by Schirmer's test, ocular surface inflammation assessed by tear matrix metalloproteinase-9 (MMP-9), corneal topography, optical biometry parameters, meibomian gland function, and patient-reported discomfort related to eye drop use.

Clinical assessments will be conducted at baseline, on the day of surgery, and at postoperative follow-up visits according to the study schedule. Safety will be monitored throughout the study by assessing adverse events and ocular findings at each visit.

This study aims to determine whether rebamipide is non-inferior to diquafosol in maintaining tear film stability and improving dry eye symptoms during the perioperative period of cataract surgery, thereby providing evidence to guide optimal dry eye management strategies in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 40 years or older scheduled for unilateral cataract surgery
* Presence of dry eye disease, defined by an Ocular Surface Disease Index (OSDI) score ≥12 and at least one of the following:

  * Tear film breakup time (TBUT) ≤7 seconds
  * Oxford corneal staining grade ≥1
  * Schirmer's test value ≤10 mm/5 minutes
* Ability and willingness to comply with the study protocol and follow-up schedule
* Provision of written informed consent

Exclusion Criteria:

* Active ocular infection or inflammation, including infectious keratitis
* History of ocular surgery other than cataract surgery in the study eye
* Use of topical medications that may affect the ocular surface (e.g., intraocular pressure-lowering eye drops)
* Any ocular or systemic condition judged by the investigator to interfere with study participation or outcome assessment

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Change in Tear Film Breakup Time (TBUT) | From baseline to postoperative 1 month
  Change in tear film breakup time (TBUT) from baseline to the postoperative period, comparing rebamipide and diquafosol for perioperative management of dry eye disease in patients undergoing cataract surgery.

SECONDARY OUTCOMES:
Change in Ocular Surface Disease Index (OSDI) Score | From baseline to postoperative 1 and 3 months
  Change in patient-reported dry eye symptoms assessed using the Ocular Surface Disease Index (OSDI) questionnaire.
Change in Corneal Staining Grade (Oxford Scale) | From baseline to postoperative 1 month
  Change in corneal epithelial staining graded using the Oxford scale following fluorescein staining.
Change in Schirmer's Test Value | From baseline to postoperative 1 and 3 months
  Change in tear secretion measured by Schirmer's test without anesthesia.
Change in Tear Matrix Metalloproteinase-9 (MMP-9) Level | From baseline to postoperative 1 and 3 months
  Change in tear matrix metalloproteinase-9 (MMP-9) levels assessed using a commercially available tear MMP-9 test.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Mec, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
The detailed study protocol and the data that support the findings of this study are available from the corresponding author upon reasonable request.